CLINICAL TRIAL: NCT01609114
Title: Irradiation Modulates the Pharmacokinetics of Anticancer Drugs for Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH No.:100163-F
Record Dates: First submitted 2012-04-27; First posted 2012-05-31 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Head and Neck Cancer
Keywords: phenomena and mechanism of RT-PK; fact for different anticancer drugs; different part in human
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control groups: chemotherapy (C/T) is applied in the morning. After 4-6 hrs, RT is delivered (according to the clinical practice).
- experimental groups: RT is delivered in the morning. After 4-6 hrs, C/T is applied.

SUMMARY:
The concurrent use of chemotherapy during radiation therapy (CCRT) is now the important treatment stratagem for locally advanced head and neck cancer or nasopharyngeal cancer (NPC). For these cases, 5-Fluorouracil (5-FU) and cisplatin (CDDP) are the most commonly used agents of CCRT. It plays an important role to improve the treatment outcome and increases the opportunities for organ preservation.

In the past, Radiotherapy (RT) was solely used as a local treatment and its effect was estimated by local effect model. However, growing evidence shows that irradiation has direct DNA damage-dependent effects as well as sending signals to neighboring cells. Recently, the investigators reported that abdominal irradiation could significantly modulate the systemic pharmacokinetics of 5-FU at 0.5 Gy, off-target area in clinical practice, and at 2 Gy, the daily treatment dose for target treatment in an experimental rat model. Additionally, the results from a clinical investigation showed that colorectal cancer patients with lower AUC of 5-FU during adjuvant chemotherapy had lower disease-free survival. Taken together, these lines of evidence support the importance and necessity to search for the mediators responsible for the unexpected effect of local RT on systemic pharmacokinetics of chemotherapeutic agents, such as 5-FU.

In the present study, the investigators examined whether the phenomena and mechanism of RT-PK(pharmacokinetics) is a fact for different anticancer drugs and for different part in human.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced head and neck, nasopharyngeal cancers, who prepares for concurrent chemoradiation therapy as definitive or adjuvant setting

Exclusion Criteria:

* previous cancer history；abnormal function of liver and kidney, immunol disease or hematologic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chemotherapy-naive patients with histologically confirmed, locally advanced head and neck, nasopharyngeal cancers, who prepares for concurrent chemoradiation therapy as definitive or adjuvant setting, are consecutively enrolled in this study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of'chemo-drugs" | "15, 30, 45, 60, 90, 120 min post-dose"

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan, Taiwan

REFERENCES:
- [Derived] Hsieh CH, Hou ML, Chiang MH, Tai HC, Tien HJ, Wang LY, Tsai TH, Chen YJ. Head and neck irradiation modulates pharmacokinetics of 5-fluorouracil and cisplatin. J Transl Med. 2013 Sep 26;11:231. doi: 10.1186/1479-5876-11-231. PMID 24066670